CLINICAL TRIAL: NCT04607694
Title: DAHANCA 35: A Randomized Trial of Proton Versus Photon Radiotherapy for the Treatment of Head-neck Cancer
Brief Title: DAHANCA 35: Proton Versus Photon Therapy for Head-neck Cancer
Acronym: DAHANCA 35
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Head and Neck Cancer Group (Network)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAHANCA 35
Record Dates: First submitted 2020-10-19; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Head-and-neck Cancer
Keywords: Proton radiotherapy; DAHANCA
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proton radiotherapy (Experimental): Proton radiotherapy according to the guidelines defined by the Danish Head-Neck Cancer Group (DAHANCA). Treatment: 66-68 Gy/ 33-34 fx/ 6/W, with cisplatin 40 mg/m2/W and nimorazole to suitable patients
  Interventions: Radiation: Proton radiotherapy
- Photon radiotherapy (Active Comparator): Photon radiotherapy according to the guidelines defined by the Danish Head-Neck Cancer Group (DAHANCA). Treatment: 66-68 Gy/ 33-34 fx/ 6/W, with cisplatin 40 mg/m2/W and nimorazole to suitable patients
  Interventions: Radiation: Photon radiotherapy

INTERVENTIONS:
Radiation: Proton radiotherapy — Proton radiotherapy
  Arms: Proton radiotherapy
Radiation: Photon radiotherapy — Photon radiotherapy
  Arms: Photon radiotherapy

SUMMARY:
Patients with squamous cell carcinoma of the pharynx or larynx and an anticipated benefit of proton radiotherapy in reducing the risk of late dysphagia or xerostomia are randomized to proton or photon radiotherapy (2:1)

DETAILED DESCRIPTION:
DAHANCA 35 is two parallel conducted, but separate randomized studies, within the same trial (DAHANCA 35D and DAHANCA 35X) by the Danish Head-Neck Cancer Study Group (DAHANCA). In patients with squamous cell carcinoma of the pharynx or larynx planned for primary radiotherapy a proton and a photon doseplan is prepared. If proton radiotherapy reduces the anticipated absolute risk of dysphagia >= grade 2 (DAHANCA scale, DAHANCA 35D) or severe xerostomia >= grade 4 (EORTC Head-Neck 35, DAHANCA 35X) more than 5%, the patient is randomised to either proton therapy or photon therapy, 2:1. The anticipated risk of xerostomia and dysphagia is estimated using Normal-Tissue Complication Models (NTCP). Patient are analysed according to the primary endpoint (dysphagia and/or xerostomia) after which they were enrolled. DAHANCA 35D is expected to enroll 360 patients and DAHANCA 35X 240 patients (in total 600 patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven squamous cell carcinoma of the pharynx or larynx planned for primary radiotherapy with curative intent
* A predicted clinical significant reduction in the risk of any of the two primary endpoints (>= grade 2 observer-rated dysphagia or grade 4 patient-reported xerostomia) after proton therapy compared to photon therapy based on comparison of the individual patient dose plans
* No current or earlier malignancies, which may influence treatment, evaluation or outcome of the head-neck cancer
* Informed consent as required by law
* Above 18 years of age

Exclusion Criteria:

* Patient with cancers of the glottic larynx (stage I/II), skull base, sino-nasal area, unknown primary tumor and prior malignancies.
* Patients with contraindications for proton therapy. Per October 2020, this includes pacemakers, implanted defibrillators and tracheostomy
* Inability to attend full course of radiotherapy or follow-up visits in the outpatient clinic
* Distant metastasis
* Previous radiotherapy of the head and neck
* Previous surgery for the primary cancer with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Dysphagia >= grade 2 | Six months after end of radiotherapy
  The rate of observer-reported dysphagia >= grade 2 measured by the DAHANCA late toxicity score (grade 0-4, with 0 being best)
Xerostomia = grade 4 | Six months after end of radiotherapy
  The rate of patient-reported xerostomia measured by the EORTC Quality of life questionnaire (QLQ) Head-Neck (HN) 35 (grade 1-4, with 1 being best)

SECONDARY OUTCOMES:
Loco-regional tumor control | Up to five years after end of radiotherapy
  Time to event of local-regional failure, from date of randomization to the date of first documented loco-regional failure. Rates are estimated by the Kaplan-Meier method. Interim analyses after 100, 200 and 300 patients. Will not be reported before the primary endpoint.
Overall survival | Up to five years after end of radiotherapy
  From date of randomisation to date of death
Number of participants with disease-free survival | Up to five years after end of radiotherapy
  From date of randomization to date of death (all causes), loco-regional failure or distant failure, whichever comes first
Disease-specific survival | Up to five years after end of radiotherapy
  From date of randomization to date of death (by loco-regional or distant failure)
Acute toxicity | From the beginning of and up to two months after end of radiotherapy
  DAHANCA acute toxicity score (grade 0-4, 0 being best)
Late toxicity | From two months to five years after end of radiotherapy
  DAHANCA late toxicity score (grade 0-4, 0 being best)
EORTC QLQ-Head-Neck 35 | Up to ten years after end of radiotherapy
  Swallowing and social-eating scale and specific HN35 items related to eating and pain (grade 1-4, 1 being best)
EORTC C30 | Up to ten years after end of radiotherapy
  Specific C30 items related to fatigue, nausea and vomiting (grade 1-4, 1 being best)
MD Anderson Dysphagia Index | Up to ten years after end of radiotherapy
  MD Anderson Dysphagia Index (MDADI) (grade 1-5, 1 being best)
EuroQol Five Dimension Scale (EQ-5D) | Up to ten years after end of radiotherapy
  Quality-adjusted life-years
Composite time corrected toxicity score (CTCT) | Up to five years after end of radiotherapy
  The sum of the time corrected dysphagia score and the time corrected xerostomia score normalised to maximum score across all days using EORTC QLQ-Head-Neck 35. The measure is unit-less.
Modified barium swallowing | One year after end of radiotherapy
  Functional swallowing test - DIGEST scale (grade 0-4, 0 being best)
Stimulated whole-mouth salivary flow | Up to five years after end of radiotherapy
  Stimulated whole-mouth salivary flow

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Friborg, MD, PhD, Principal Investigator — Danish Head-Neck Cancer Group (DAHANCA)
Locations (7):
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Danish Center for Particle Therapy, Aarhus
  - Herlev Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Næstved Hospital, Næstved
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No